CLINICAL TRIAL: NCT01561443
Title: LINE: Treatment Patterns in postmenopausaL Women With Hormone Receptor Positive Breast Cancer
Acronym: LINE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ORU-XXX-2011/1
Record Dates: First submitted 2012-03-19; First posted 2012-03-23 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Local Advanced or Metastatic Postmenopausal Breast Cancer
Keywords: Breast cancer,; hormone positive,
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is the first study focused on features/stereotypes of the first and second-line treatment patterns in Russia, comparison of different treatments, and determination of effective hormone treatment patterns in real-life practice with evaluation of pharmacoeconomic aspects. Study LINE is designed for collection of data on clinical effectiveness of second-line hormone treatment and quality of life in patients with breast cancer(BC).

DETAILED DESCRIPTION:
LINE: Treatment patterns in postmenopausaL women wIth hormone receptor positive breast caNcEr

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with hormone receptor-positive breast cancer:
* Recurrence after the adjuvant hormone therapy;
* Or initially inoperable locally advanced or metastatic breast cancer progressed after the first line hormone therapy;
* Ability to read and write and complete questionnaires Provision of written informed consent
* Patients who have already been prescribed therapy with the above-mentioned lines and who can continue on the prescribed therapy in the investigator's opinion according to his/her regular clinical practice and cure

Exclusion Criteria:

* As per study design, to ensure high validity of data and to obtain accurate information on real-life practice,
* Patients currently participating in other clinical studies will not be included in this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hormone positive, postmenopausal breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Collection of data of routine regimens of hormone therapy in postmenopausal women with hormone receptor-positive, locally advanced or metastatic breast cancer | 2 years

SECONDARY OUTCOMES:
Quality of life (QoL): the extent of reduction in QoL deficit from 1 visit | 2 years
The extent of reduction anxiety inventory | 2 years
Effectiveness: Tumor regression; number of patients with complete response (CR), partial response (PR) or stable disease | 2 years
Historical data analysis: treatment patterns effectiveness, duration of the adjuvant or first-line hormone treatment | 2 years
Response duration | 2 years
Performance status (ECOG) | 2 years
Co-morbidities and relevant historical data | 2 years
The information on spontaneous office visit to oncologist or hospitalization including reasons, diagnosis, days of hospitalization, procedures and concomitant medication changes will be collected. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Stepanov, Prof., Study Director — AstraZeneca; Maria Konstantinova, Prof, Principal Investigator — Russian Oncology Scientific Center; Sergey Gutorov, Prof., Principal Investigator — Russian Oncology Scientific Center; Marina Stenina, PhD, Principal Investigator — Surgery Institute named after A.V. Vishnevskiy
Locations (19):
- Russia (19):
  - Research Site, Chita
  - Research Site, Irkutsk
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Khanty-Mansiysk
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Perm
  - Research Site, S-Petersburg
  - Research Site, Samara
  - Research Site, Tula
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Vladivostok
  - Research Site, Volgograd
  - Research Site, Yaroslavl

REFERENCES:
- See also: Clinical study report synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1020&filename=NIS-ORU-XXX-2011-1_Final_Report_Synopsis.pdf
- See also: CSR_synopis_NIS-ORU-XXX-2011/1 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1020&filename=NIS-ORU-XXX-2011_1_Final_Report_Synopsis.pdf